CLINICAL TRIAL: NCT06722872
Title: Effect of Laughter Therapy on Psychological Well-being, Life Satisfaction and Mental Health of the Elderly Living in a Nursing Home
Brief Title: The Effect of Laughter Therapy on the Mental Health of Elderly Living in a Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Özge Karaca, Research Asisstant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstanbulUC-NURS-OK-01
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Laughter; Mental Health Issue; Life Satisfaction; Well-Being, Psychological; Elderly
Keywords: Laughter therapy; Old age; Psychological well-being; Life satisfaction; Mental health
MeSH Terms: conditions — Laughter; Personal Satisfaction; Psychological Well-Being | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with experimental and control groups
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to prevent selection bias in the study, the assignment to the experimental and control groups will be made on a computer by a person who is unfamiliar with the research process. Individuals included in the study will not be told whether they are in the experimental or control group. The analysis of the data will be done by a statistics expert who is outside the research process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter therapy group (Experimental): Pre-tests were collected 10 days before the therapy began. The elderly participants were introduced individually and informed face-to-face about laughter therapy. Therapy sessions were conducted face-to-face twice a week, with a total of 12 sessions. Each laughter therapy session lasted 50 minutes. Post-tests were collected immediately after the final therapy session. Four weeks later, follow-up tests were also conducted face-to-face.
  Interventions: Other: Laughter therapy
- No intervention group (No Intervention): The control group did not receive laughter therapy; they continued with routine nursing home care. Pre-tests, post-tests, and follow-up tests were collected on the same days as the experimental group. After the follow-up tests were completed, a 30-minute laughter therapy session was provided to control group participants who wished to participate.

INTERVENTIONS:
Other: Laughter therapy — Laughter therapy, developed by Dr. Madan Kataria in 1995, is a structured exercise program use of laughter and breathing exercises.Laughter therapy sessions begin with warm-up techniques, including clapping, singing, and stretching movements. These are followed by breathing exercises to prepare the lungs for laughter. After the breathing exercises, laughter is simulated using acting techniques. Shortly thereafter, the simulated laughter spreads from person to person through group dynamics, transforming into genuine laughter, which is then followed by a series of laughter exercises. A laughter therapy session may conclude with laughter meditation, during which participants allow natural laughter to flow freely, followed by guided relaxation exercises. To maximize the benefits of laughter's contagious nature, it is recommended that laughter therapy be conducted in groups. Each session varies depending on the target audience, typically lasting around 45 minutes.
  Arms: Laughter therapy group

SUMMARY:
This study was designed and conducted as a randomized controlled experimental research with a pre-test and post-test control group to evaluate the effect of laughter therapy on psychological well-being, life satisfaction, and mental health of elderly individuals living in a nursing home.

DETAILED DESCRIPTION:
Among the most important indicators of successful aging are individuals' ability to derive satisfaction from life, maintain cognitive and social competence, sustain mental and physical health, possess a sense of personal control, and experience increased longevity. Supporting elderly individuals to live independently, maintaining their social relationships, and encouraging healthy lifestyle behaviors are key to achieving an active and successful aging process.

Life satisfaction is considered one of the most significant factors influencing mental health and determining adaptation during all stages of life, particularly in old age. As an indicator of well-being, life satisfaction has a positive correlation with psychological resilience and mental health. Thus, psychological well-being, life satisfaction, and mental health of elderly individuals are interconnected, and interventions aimed at enhancing well-being and life satisfaction are known to positively affect the mental health of older adults.

In this context, laughter therapy has recently gained attention as an approach with observed positive effects on the physical and mental health of elderly individuals. Laughter therapy, developed by Dr. Madan Kataria in 1995, aims to support physical and mental health through laughter and breathing exercises.

Meta-analyses and systematic reviews indicate that laughter therapy has positive psychosocial effects on older adults, including reducing depression, perceived stress, and anxiety, enhancing psychological well-being, regulating blood pressure and cortisol levels, improving sleep and quality of life, reducing death anxiety, loneliness, and depressive tendencies, and increasing happiness, life satisfaction, and mood. Laughter therapy is considered a non-invasive, non-pharmacological, cost-effective, accessible, and easy-to-apply complementary/alternative therapy, with calls for further evidence-based studies to promote its use.

Within this framework, the aim of this research is to determine the effect of laughter therapy on the psychological well-being, life satisfaction, and mental health of elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 65
* Scoring ≥ 18 points on the Mini-Mental Examination
* Having the ability to communicate
* Not having participated in a laughter therapy session before

Exclusion Criteria:

* Having severe hearing or perception impairment that hinders communication
* Having a physical or psychological condition that prevents participation in therapy
* Having moderate-to-severe Alzheimer's disease, uncontrolled hypertension, epilepsy, abdominal surgery within the past 3 months, or a surgical procedure with a risk of bleeding
* Choosing not to continue participating in the study

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being Scale for Older Adults | Pre-test, Post-test (6th week), Follow-up Test (4th week)
  The scale was used to measure the psychological well-being levels of older adults. It consists of 15 items in a 5-point Likert format (1 = Strongly Disagree to 5 = Strongly Agree). No specific cutoff score has been determined for the well-being levels of older adults. Higher scores indicate an increase in the level of well-being. The minimum score obtainable from the scale is 15, while the maximum score is 75.
Life Satisfaction Scale for Older Adults | Pre-test, Post-test (6th week), Follow-up Test (4th week)
  The scale was used to assess the participation of older adults in the process of life satisfaction. It consists of 14 items across 3 subdimensions and is structured as a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree). The scale includes 9 items under the "Self-Acceptance" subdimension, 2 items under the "Motivation" subdimension, and 3 items under the "Peace" subdimension. Scores range from 14 to 70, with individual subdimension scores calculated by dividing the total score by the number of items in each subdimension. The "Self-Acceptance" subdimension ranges from 9 to 45, the "Motivation" subdimension from 2 to 10, and the "Peace" subdimension from 3 to 15.
Depression Anxiety Stress Scale (DASS-21) | Pre-test, Post-test (6th week), Follow-up Test (4th week)
  The scale was used to assess the mood of older adults by identifying their levels of depression, anxiety, and stress. DASS-21 is a shortened version of the 42-item Depression Anxiety Stress Scale. It consists of 21 items in a 4-point Likert format (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always) and includes three subdimensions: depression, anxiety, and stress. Each subdimension is measured by 7 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- KASEV Huzurevi, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No